CLINICAL TRIAL: NCT01141881
Title: Evaluation of the Role of Intravitreal Injection of TPA in Treatment of Refractory Diabetic Macular Edema
Brief Title: Evaluation of the Role of Intravitreal Tissue Plasminogen Activator in Treatment of Refractory Diabetic Macular Edema
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: occurrence of retinal hemorrhage , increase in macular edema of some patients in TPA group
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: naser shoeibi, Professor assistant of ophthalmology
Masking: Single | Purpose: Treatment
Other Study IDs: 2202
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2008-09

CONDITIONS: Diabetic Macular Edema
Keywords: Tissue Plasminogen activator,; Clinically significant macular edema,; Refractory Diabetic macular edema ,; posterior vitreous detachment
MeSH Terms: conditions — Vitreous Detachment | interventions — Tissue Plasminogen Activator; Bevacizumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TPA,IVB,F/U (Experimental)
  Interventions: Drug: Tissue Plasminogen Activator,bevacizumab ,follow up

INTERVENTIONS:
Drug: Tissue Plasminogen Activator,bevacizumab ,follow up — 25 microgram in 0.05 cc,1.25 mg in 0.05 cc,nothing
  Other Names: bevacizumab :avastin

SUMMARY:
Purpose: to evaluate the effect of intravitreal injection of tissue plasminogen activator(tPA) in treatment of refractory diabetic macular edema(DME).

ELIGIBILITY:
Inclusion Criteria:

1. type 2 diabetes
2. Non proliferative diabetic retinopathy(NPDR) stage of diabetic retinopathy
3. patients with refractory DME CSME (patients with the last MPC at least 3 months before and no improvement was observed in BCVA, macular thickness inOCT, clinical examination and fundus photographs of patients )
4. Absence of PVD in the B-scan
5. Absence of PVD in OCT of macular area and optic disk
6. Absence of PVD in slit lamp biomicroscopy(SLE)
7. the last PRP session was at least 3 months ago.
8. Absence of traction on macula in clinical examination and OCT

Exclusion Criteria:

1. One eye patients
2. Patients who are candidates for intraocular surgery.
3. Patients with the history of glaucoma or ocular hypertension
4. Patients with a history of vitrectomy in the study eye
5. Not being able to refer for the next visits
6. Eyes with cataract that makes the assessment of the macula impossible.
7. Intraretinal hemorrhage at fovea that will interfere with OCT.
8. BCVA ≤ 0.1

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2009-05; Primary Completion 2010-01 (Estimated); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: naser shoeibi, MD, Study Director — mashhad university of medical science
Locations (1):
- Khatam Hospital, Mashhad, Khorasan Razavi, Iran

REFERENCES:
- [Background] Murakami T, Takagi H, Ohashi H, Kita M, Nishiwaki H, Miyamoto K, Watanabe D, Sakamoto A, Yamaike N, Yoshimura N. Role of posterior vitreous detachment induced by intravitreal tissue plasminogen activator in macular edema with central retinal vein occlusion. Retina. 2007 Oct;27(8):1031-7. doi: 10.1097/IAE.0b013e318074bc39. PMID 18040240